CLINICAL TRIAL: NCT03690830
Title: Use of Metabolomics for the Identification of Endometrial Biomarkers for Recurrent Pregnancy Loss and Reccurent Implantation Failure Following in Vitro Fertilization.
Brief Title: Use of Metabolomics for the Identification of Endometrial Biomarkers for IRPL and RIF After in Vitro Fertilization
Acronym: ENDOMETAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RCB n°2018-A01871-54
Record Dates: First submitted 2018-09-17; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Recurrent Pregnancy Loss; Recurrent Implantation Failure
Keywords: Metabolomic; Endometrial biomarkers; Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Two case groups (Recurrent Implantation Failure and idiopathic recurrent pregnancy loss ) One control group (patients undergoing Assisted ReproductiveTechnologies (ART) for male factor infertility)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Case group RIF (Experimental): blood samples, analyzing endometrial cells
  Interventions: Other: metabolomics analysis
- Case group IRPL (Experimental): blood samples, analyzing endometrial cells
  Interventions: Other: metabolomics analysis
- Control group (Active Comparator): blood samples, analyzing endometrial cells
  Interventions: Other: metabolomics analysis

INTERVENTIONS:
Other: metabolomics analysis — collect blood samples and endometrial cells

SUMMARY:
It is a case-control study composed of 3 groups : 2 cases groups (RIF and IRPL) already composed as part of a pre-existing research project and 1 control group including patients undergoing ART for male factor infertility.

The purpose of this study is to compare the 2 case group with the control group to identify metabolomics signatures.

DETAILED DESCRIPTION:
The investigators have designed a unicentric, case-control, retro- and prospective study to compare the endometrial metabolomics profile in three groups of patients. The two case groups (RIF and IRPL) are already composed and the endometrial and blood samples already taken as part of a pre-existing research project. The current protocol concerns the control group that includes patients undergoing ART for male factor infertility.

The study will include three groups. The first group is composed of patients with a history of RIF following IVF-ET. RIF is defined as failure to obtain a clinical pregnancy (fetal cardiac activity at 6-7 weeks gestational age (GA)) following at least 3 different transfers of at least 4 good quality embryos (fresh or frozen).

The second group comprises patients with a history of IRPL, defined as three or more consecutive pregnancy losses that occurred before 14 weeks gestational age. Early pregnancy losses diagnosed before ultrasonographic confirmation will be included.

The third group will include patients undergoing ART for male factor infertility.

The study protocol will be presented and explained to all eligible patients in the control group during the routine consultation before treatment. Patients who agree to participate will contact the department to program the inclusion visit with one of the attending physicians in the department, during which the blood and endometrial samples will be taken. The inclusion visit will take place at the department of reproductive medicine of Angers University Hospital around day 21 of the menstrual cycle (in the middle of the implantation window, which occurs between day 19 and 23 of the cycle, day 1 being the first menstruation day).

The metabolomics analysis will be performed according to the same protocol for all samples (study and control groups)

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 (included) and 40 years (excluded).
* Patients who agreed to participate and signed the consent form
* Patients undergoing ART for male factor infertility: male partner with severe oligoasthenospermia or azoospermia.
* Patients without any prior history of infertility or risk factors for infertility other than the male factor.
* Patients with a normal basic infertility workup prior to ART (Day 3 serum FSH, LH, Estradiol and AMH; Antral follicle count; hysterosonography or hysterosalpingography)

Exclusion Criteria:

* Non-French speaking patients.
* Major patients that are wards of the nation.

  * Patients deprived of their liberty on criminal charges or for civil reasons.
  * Patients under psychiatric care.
  * Patients under legal protection.
  * Patients unable to sign consent forms.
* Patients not covered by social security (which covers all treatments administered).
* Patients currently participating in other interventional research projects.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women pregnancy
Enrollment: 40 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Analyze the endometrial samples with mass spectrometry using the Biocrates kit (measures 188 metabolites) | 1 day
  To compare the metabolomics profile of the endometrium in patients with RIF or IRPL following IVF-ET to patients undergoing Assisted Reproductive Technologies (ART) for male factor infertility to see if there is any significant difference, qualitative or quantitative or both in the metabolites.

SECONDARY OUTCOMES:
Analyze the blood sample with standard biological examination and the endometrial sample with mass spectrometry using the Biocrates kit | 1 day
  To compare the metabolomics profiles based on endometrial cells to profiles based on blood samples, and to compare the profiles between the 2 groups (RIF and IRPL). If any difference, analyze the mecanisms behind it.
Analyze the endometrial samples with mass spectrometry using the Biocrates kit | 1 day
  To analyze the endometrial metabolomics profile according to the etiology of infertility in the group of patients with RIF following IVF-ET (endometriosis, low ovarian reserve, polycystic ovarian syndrome…).

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University hospital, Angers, Maine Et Loire, France

IPD SHARING:
Plan to Share IPD: Yes